CLINICAL TRIAL: NCT06938217
Title: Safety and Efficacy of Low-Flow ECMO in a Multi-modal Cohort of Adults in Respiratory Failure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Extracorporeal Life Support (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, Jeffrey DellaVolpe, Medical Director, Institute for Extracorporeal Life Support; Intensivist, Institute for Extracorporeal Life Support
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LFECMO-01
Record Dates: First submitted 2025-01-28; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Hypoxemic Respiratory Failure; Mechanical Ventilation; Acute Respiratory Distress Syndrome (ARDS)
Keywords: Extracorporeal Life Support; Low-Flow ECLS; Mechanical Ventilation; Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Initiation of low-flow ECLS (Other): To evaluate the safety, feasibility, and efficacy of low-flow ECLS and assess the feasibility of its use
  Interventions: Device: Low-flow ECMO

INTERVENTIONS:
Device: Low-flow ECMO — low-flow ECMO, defined as 1-2.5 L of blood flow/min.

SUMMARY:
The current standard of care (SOC) for treatment of patients with acute respiratory distress syndrome (ARDS), inhalation injury, volume overload, and/or pulmonary dysfunction is mechanical ventilation (MV). However, these techniques are associated with several complications after prolonged use, including risk of infection, increased sedation requirements, pulmonary edema, ventilator-induced lung injury (VILI), barotrauma, and multi-organ failure.

Extracorporeal life support (ECLS) has been used to successfully minimize, replace, or avoid the use of MV. This concept is critical as it permits ultra-lung protective MV settings, mobilization, early ambulation of patients, and timely extubation (when appropriate).

Conventional ECLS typically requires blood flows of 3-6 L/min, and its cannula sizes range from 21-25 Fr. This is by definition "high-flow" as it constitutes near-complete extracorporeal circulation of patient's circulating blood volume. On the other hand, low-flow ECLS at 1-2.5 L/min has been shown to prevent deleterious shifts in pH and PaCO2 at a lower level of invasiveness, and its cannula sizes range from 19-20 Fr dual lumen cannulas (which are associated with less serial dilation). The investigators propose the use of a low-flow circuit to include the NovaLung system in conjunction with a smaller tubing set and cannula to enable earlier utilization of ECLS with less invasiveness and smaller catheters. Specifically, the study will either utilize the Crescent RA cannula (or equivalent dual-lumen cannula) or use a 15-25 Fr cannula, both with 3/8 tubing/step-down tubing, as needed, for our study. A femoral (fem)-femoral or femoral-internal jugular (IJ) approach may also be used.

Carbon dioxide is six times more diffusible than oxygen across the membrane; thus, carbon dioxide transfers can occur with high efficiency at our targeted blood flows of 1-2.5L/min. Oxygen can still transfer at these blood flows, and low flow can improve oxygen levels to some degree.

There are three benchtop-based manuscripts that suggest that low-flow ECMO is associated with a potential increase in factors that increase the risk of bleeding complications/circuit changes. However, the manuscripts either tested <1 L/min blood flow rates, or the effect of cannula size was not considered. None of them included the biological component of endothelial interaction. Mitigating the risk of bleeding complications by will be completed by administering anticoagulants with a target PTT of 40-50 seconds, and by monitoring the patients and their coagulation panels closely. There may be less risk of circuit clotting in our study because of chosen flow rates (1-2.5 L/min).

DETAILED DESCRIPTION:
The investigators focus is to demonstrate the safety, feasibility, and efficacy of low-flow ECLS as a treatment for multiple respiratory conditions (including ARDS, volume overload, obstructive and restrictive pulmonary diseases, hypoxia) in conjunction with MV.

BACKGROUND

The two most significant trials in the last five years investigating strategies around low-flow ECLS with the intent of CO2 reduction/ventilator reduction are as follows:

* SUPERNOVA Multi-Center Phase II Study in Europe and Canada: In 2019 Combes et al assessed the feasibility and safety of lower CO2 extraction ECLS devices (300-500 mL/min) in patients with moderate ARDS compared to higher CO2 extraction ECLS devices (800-1000 mL/min, N=95). The authors concluded that the use of low-flow ECLS to facilitate ultra-protective ventilation was feasible, and that it mitigated respiratory acidosis in patients with moderate ARDS.
* REST Multi-Center Randomized Clinical Trial (RCT) in the United Kingdom: In 2021 McNamee et al set to determine whether lower tidal volume MV using extracorporeal CO2 removal improves outcomes in adult patients with acute hypoxemia respiratory failure (n=202) compared to conventional low tidal volume MV (n=210). There were significantly fewer mean ventilator-free days in the extracorporeal CO2 removal group compared with the SOC (p=0.02). However, the trial was halted because of futility and feasibility. Although the conclusion was that the use of extracorporeal CO2 removal did not significantly reduce 90-day mortality (p=0.68), the study may have been underpowered to detect an important difference. Furthermore, the most notable limitation of the study was that the duration of low-flow ECLS was limited to less than 7 days (which caused discontinuation of the intervention in 33 patients). The authors state that "it is possible that a longer duration of ECCO2R with greater tidal volume reduction may have been required to demonstrate an effect because higher intensities of invasive MV have been shown to be associated with increased risk of death in a time-dependent fashion". Additional limitations of the study were that (1) only 6% of the screened patients were included in the study, (2) 8% of the randomized subjects in the intervention group did not receive the intervention, and (3) most of the sites had not performed ECLS before the initiation of the study, leading to practical inexperience potentially negatively influencing the outcomes of the intervention group.

The investigators note several differences in their protocol that differentiates it from the REST trial. First, the investigators will use a device capable of obtaining higher blood flow rates with higher initial targets of blood flow (1-2.5L/minute). Specifically, the study will use a low-flow circuit to include the NovaLung system (Fresenius Medical Care, Waltham MA) in conjunction with a smaller tubing set and cannula (15 - 25 Fr versus 23 - 31 for conventional ECMO, as needed) to enable earlier utilization of ECLS with less invasiveness and smaller catheters. Second, the current study includes broader limitations to length of time of the device (e.g. 28 days versus 7 days), which may be a more pragmatic and generalizable approach.

RATIONALE The current standard of care (SOC) for treatment of patients with acute respiratory distress syndrome (ARDS), inhalation injury, volume overload, and/or pulmonary dysfunction is mechanical ventilation (MV). However, these techniques are associated with several complications after prolonged use, including risk of infection, increased sedation requirements, pulmonary edema, ventilator-induced lung injury (VILI), barotrauma, and multi-organ failure. Extracorporeal life support (ECLS) has been used to successfully minimize, replace, or avoid the use of MV. This concept is critical as it permits ultra-lung protective MV settings, mobilization, early ambulation of patients, and timely extubation (when appropriate).

Low-flow ECLS has been shown to prevent deleterious shifts in pH and PaCO2 at a lower level of invasiveness. The investigators hypothesize that the use of low-flow ECLS will be a safe option for the treatment of pulmonary dysfunction and mild and moderate ARDS, that it will significantly reduce MV settings, and that it will decrease the need for intubation for patients requiring respiratory support for either failure to oxygenate or ventilate.

PROCEDURES Subjects meeting criteria for enrollment will be screened by the Principal Investigator or any delegates assigned to review the patient's chart. A HIPAA authorization and informed consent will be provided by the subject or legally authorized representative (LAR) prior to conducting any additional research procedures.

Patients enrolled after consent is obtained will be placed on Low-Flow ECMO by trained physicians. Subjects will be cannulated in one of two ways, either at bedside with the use of radiographic imaging to confirm accurate cannula placement, or in the catheter laboratory under fluoroscopy with safety measures in place to appropriately monitor the patient's vital signs, ventilatory measurements, and LF ECMO settings.

Initiation of LF ECMO will require cannula placement and connection to the Novalung XLung extracorporeal circuit. Size and type of cannula will be determined by the investigator and documented at cannulation. The XLung will be used with circuit to accommodate lower flows necessary to efficiently move 1-2.5 LPM of blood through the oxygenator. Subjects treated with low-flow ECMO will receive systemic anticoagulation per standard of care for patients treated with ECLS. After cannulation and placement on LF ECMO, blood gases will be drawn from the patient, pre-Xlung, and post-Xlung to assess the function of the Novalung system, patient's stability after initiation, and the ability to effectively wean ventilatory support.

Multiple labs will be collected and documented as routine standard of care while others will be collected prior to device implementation and during the duration of therapy for research purposes. The following is considered standard of care (as needed, daily): arterial blood gases, lactate, platelet count. Standard of care costs are billed to insurance. The following are considered research costs (prior to device initiation, within one hour of device initiation [if collected]): arterial blood gases, lactate, platelet count. Heparin doses, aPTT, ACT, anti-Xa, plasma-free hemoglobin, pre- and post-membrane analyses are all research costs, in addition to inflammatory markers and functional outcomes (6MWT, quality of life questionnaires). All research costs are covered by the awarded grant.

Biospecimens: Approximately 2 mLs of blood will be collected in tubes containing EDTA at least seven times (pre-ECLS, daily, post-ECLS, discharge, 30-, 60-, 90-days post-discharge, as available). Blood will be taken prior to the administration of anesthesia (when applicable), from an existing catheter, or by venipuncture. The samples will be placed on ice, and blood will be separated by centrifugation within 30 minutes of collection to yield roughly 1 mL of plasma. The samples will be stored in appropriate freezer (long-term of ≤-80ºC or temporarily ≤-20°C). Urine (up to 10 mLs) will be collected either from the subject's urinary retention catheter or directly from the subject in a urine cup, and it will be stored in appropriate freezer (long-term of ≤ -80ºC or temporarily ≤ -20°C) until analysis.

ELIGIBILITY:
Inclusion Criteria

Acute hypoxemic respiratory failure meeting all the following criteria:

* New or worsening respiratory symptoms developing within 2 weeks prior to the onset of need for oxygen or respiratory support
* Endotracheal mechanical ventilation for ≤ 5 days
* PaO2/FiO2 ≤ 200 mmHg for at least 6 hours, or for at least two readings one hour apart
* Male or non-pregnant female
* Admitted to the ICU at MHS
* Age ≥ 18 years

Exclusion Criteria

* Hypoxemia is primarily attributable to fluid overload from acute heart failure
* Hypoxemia is primarily attributable to pulmonary embolism
* Hypoxemia is primarily attributable to status asthmaticus
* Extubation is planned or anticipated on the day of screening
* ICU discharge is planned or anticipated on the day of screening
* The patient is moribund and deemed unlikely to survive past 24 hours (as determined by the clinical team)
* The patient has limited code status, ordered for comfort measures only, or is in hospice
* Patients over 65 years of age
* Currently receiving any form of ECLS (ex. veno-venous, veno-arterial, or hybrid configuration)
* ΔPL-dyn ≤ 20 or Static ΔP ≤ 15 cm H2O while receiving VT 6 mL/kg (i.e. normalized elastance < 2.5 cmH2O/mL/kg)
* Chronic hypercapnic respiratory failure defined as PaCO2 > 60mmHg in the outpatient setting
* Home mechanical ventilation (non-invasive ventilation or via tracheotomy), not CPAP
* Severe hypoxemia with PaO2:FiO2 < 80mmHg for >6 hours at time of screening
* Severe hypercapnic respiratory failure with pH < 7.15 and PaCO2 > 60mmHg for >6 hours at time of screening
* Expected mechanical ventilation duration < 48 hours at time of screening
* Confirmed diffuse alveolar hemorrhage from vasculitis
* Contraindications to limited anticoagulation (ex. active GI bleeding, bleeding diathesis)
* Respiratory failure known or suspected to be caused by COVID-19
* Cirrhosis of the liver (as classified stage C of the Child-Pugh Score)
* Pregnancy
* Inability to tolerate extracorporeal therapy (MAP<65 mmHg despite fluid resuscitation and vasopressors)
* Unable to obtain informed consent from either patient or legally authorized representative (LAR)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days | Documented at 28 Days
  Ventilator-free days in the first 28 days

SECONDARY OUTCOMES:
Length of Stay (LOS) | Documented at discharge from the ICU, through study completion (an average of 21 days)
  1. LOS in Intensive Care Unit (ICU)
Length of Stay (LOS) | Documented at discharge from the hospital, through study completion (an average of 21 days)
  Length of Stay in Hospital
Mortality | Documented at occurrence or death, or at discharge from the hospital, through study completion (an average of 21 days)
  In-hospital mortality
Duration | Documented daily throughout hospitalization until discharged, through study completion (an average of 21 days)
  Time to and duration of lung protective settings (Pplat≤ 28 cm H2O [protective], Pplat ≤ 25 cm H2O [ultraprotective level])
Conversion | Documented daily throughout hospitalization until discharged, through study completion (an average of 21 days)
  Conversion to full ECMO support (>2.5L/min Flow)
Adverse Events | Documented at occurrence, or daily at minimum through study completion, through study completion (an average of 21 days)
  Serious adverse events (SAEs) and Grade 3 and 4 adverse events (AEs) per Common Terminology Criteria for Adverse Events (CTCAE) v5.0 (November 2017)
Anticoagulation | Documented daily throughout hospitalization until discharged, through study completion (an average of 21 days)
  Anticoagulation (rate); results of clinical coagulation panel collected throughout hospital stay
Cardiopulmonary variables: Tidal Volume | Documented hourly and daily throughout hospitalization until discharged, through study completion (an average of 21 days)
  Tidal Volume (ml)
Cardiopulmonary variables: Minute Ventilation | Documented hourly and daily throughout hospitalization until discharged, through study completion (an average of 21 days)
  Minute Ventilation (L/min)
Cardiopulmonary variables: Respiratory Rate | Documented hourly and daily throughout hospitalization until discharged, through study completion (an average of 21 days)
  Respiratory Rate (bpm)
Cardiopulmonary variables: Heart Rate | Documented hourly and daily throughout hospitalization until discharged, through study completion (an average of 21 days)
  Heart Rate (bpm)
Cardiopulmonary variables: Arterial Blood Gas | Documented as needed for clinical care (typically Q6) throughout hospitalization until discharged, through study completion (an average of 21 days)
  Arterial Blood Gas (O2CT, O2Sat, PaO2, PaCO2, pH, HCO3)
Inflammatory Markers | Pre-ECMO, daily on ECMO, at decannulation, and at 30/60/90 day follow-up apointments
  Inflammatory markers in plasma and in urine

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D DellaVolpe, MD, MPH, Principal Investigator — Institute for Extracorporeal Life Support
Locations (1):
- Methodist Healthcare System, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzgerald M, Millar J, Blackwood B, Davies A, Brett SJ, McAuley DF, McNamee JJ. Extracorporeal carbon dioxide removal for patients with acute respiratory failure secondary to the acute respiratory distress syndrome: a systematic review. Crit Care. 2014 May 15;18(3):222. doi: 10.1186/cc13875. PMID 25033302
- [Background] Bein T, Weber-Carstens S, Goldmann A, Muller T, Staudinger T, Brederlau J, Muellenbach R, Dembinski R, Graf BM, Wewalka M, Philipp A, Wernecke KD, Lubnow M, Slutsky AS. Lower tidal volume strategy ( approximately 3 ml/kg) combined with extracorporeal CO2 removal versus 'conventional' protective ventilation (6 ml/kg) in severe ARDS: the prospective randomized Xtravent-study. Intensive Care Med. 2013 May;39(5):847-56. doi: 10.1007/s00134-012-2787-6. Epub 2013 Jan 10. PMID 23306584
- [Background] Schmidt M, Jaber S, Zogheib E, Godet T, Capellier G, Combes A. Feasibility and safety of low-flow extracorporeal CO2 removal managed with a renal replacement platform to enhance lung-protective ventilation of patients with mild-to-moderate ARDS. Crit Care. 2018 May 10;22(1):122. doi: 10.1186/s13054-018-2038-5. PMID 29743094
- [Background] Deniau B, Ricard JD, Messika J, Dreyfuss D, Gaudry S. Use of extracorporeal carbon dioxide removal (ECCO2R) in 239 intensive care units: results from a French national survey. Intensive Care Med. 2016 Apr;42(4):624-625. doi: 10.1007/s00134-016-4226-6. Epub 2016 Jan 29. No abstract available. PMID 26831671
- [Background] Ruberto F, Bergantino B, Testa MC, D'Arena C, Bernardinetti M, Diso D, De Giacomo T, Venuta F, Pugliese F. Low-flow veno-venous extracorporeal CO2 removal: first clinical experience in lung transplant recipients. Int J Artif Organs. 2014 Dec;37(12):911-7. doi: 10.5301/ijao.5000375. Epub 2015 Jan 13. PMID 25588765
- [Background] Habashi NM, Borg UR, Reynolds HN. Low blood flow extracorporeal carbon dioxide removal (ECCO2R): a review of the concept and a case report. Intensive Care Med. 1995 Jul;21(7):594-7. doi: 10.1007/BF01700166. PMID 7593903
- [Background] Ki KK, Passmore MR, Chan CHH, Malfertheiner MV, Bouquet M, Cho HJ, Suen JY, Fraser JF. Effect of ex vivo extracorporeal membrane oxygenation flow dynamics on immune response. Perfusion. 2019 Apr;34(1_suppl):5-14. doi: 10.1177/0267659119830012. PMID 30966901
- [Background] Terragni PP, Del Sorbo L, Mascia L, Urbino R, Martin EL, Birocco A, Faggiano C, Quintel M, Gattinoni L, Ranieri VM. Tidal volume lower than 6 ml/kg enhances lung protection: role of extracorporeal carbon dioxide removal. Anesthesiology. 2009 Oct;111(4):826-35. doi: 10.1097/ALN.0b013e3181b764d2. PMID 19741487
- [Background] Zochios V, Brodie D, Shekar K, Schultz MJ, Parhar KKS. Invasive mechanical ventilation in patients with acute respiratory distress syndrome receiving extracorporeal support: a narrative review of strategies to mitigate lung injury. Anaesthesia. 2022 Oct;77(10):1137-1151. doi: 10.1111/anae.15806. Epub 2022 Jul 21. PMID 35864561
- [Background] Needham DM, Colantuoni E, Mendez-Tellez PA, Dinglas VD, Sevransky JE, Dennison Himmelfarb CR, Desai SV, Shanholtz C, Brower RG, Pronovost PJ. Lung protective mechanical ventilation and two year survival in patients with acute lung injury: prospective cohort study. BMJ. 2012 Apr 5;344:e2124. doi: 10.1136/bmj.e2124. PMID 22491953
- [Background] McNamee JJ, Gillies MA, Barrett NA, Perkins GD, Tunnicliffe W, Young D, Bentley A, Harrison DA, Brodie D, Boyle AJ, Millar JE, Szakmany T, Bannard-Smith J, Tully RP, Agus A, McDowell C, Jackson C, McAuley DF; REST Investigators. Effect of Lower Tidal Volume Ventilation Facilitated by Extracorporeal Carbon Dioxide Removal vs Standard Care Ventilation on 90-Day Mortality in Patients With Acute Hypoxemic Respiratory Failure: The REST Randomized Clinical Trial. JAMA. 2021 Sep 21;326(11):1013-1023. doi: 10.1001/jama.2021.13374. PMID 34463700
- [Background] Combes A, Fanelli V, Pham T, Ranieri VM; European Society of Intensive Care Medicine Trials Group and the "Strategy of Ultra-Protective lung ventilation with Extracorporeal CO2 Removal for New-Onset moderate to severe ARDS" (SUPERNOVA) investigators. Feasibility and safety of extracorporeal CO2 removal to enhance protective ventilation in acute respiratory distress syndrome: the SUPERNOVA study. Intensive Care Med. 2019 May;45(5):592-600. doi: 10.1007/s00134-019-05567-4. Epub 2019 Feb 21. PMID 30790030
- [Background] Goligher EC, Tomlinson G, Hajage D, Wijeysundera DN, Fan E, Juni P, Brodie D, Slutsky AS, Combes A. Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome and Posterior Probability of Mortality Benefit in a Post Hoc Bayesian Analysis of a Randomized Clinical Trial. JAMA. 2018 Dec 4;320(21):2251-2259. doi: 10.1001/jama.2018.14276. PMID 30347031
- [Background] Combes A, Hajage D, Capellier G, Demoule A, Lavoue S, Guervilly C, Da Silva D, Zafrani L, Tirot P, Veber B, Maury E, Levy B, Cohen Y, Richard C, Kalfon P, Bouadma L, Mehdaoui H, Beduneau G, Lebreton G, Brochard L, Ferguson ND, Fan E, Slutsky AS, Brodie D, Mercat A; EOLIA Trial Group, REVA, and ECMONet. Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome. N Engl J Med. 2018 May 24;378(21):1965-1975. doi: 10.1056/NEJMoa1800385. PMID 29791822
- [Background] Peek GJ, Mugford M, Tiruvoipati R, Wilson A, Allen E, Thalanany MM, Hibbert CL, Truesdale A, Clemens F, Cooper N, Firmin RK, Elbourne D; CESAR trial collaboration. Efficacy and economic assessment of conventional ventilatory support versus extracorporeal membrane oxygenation for severe adult respiratory failure (CESAR): a multicentre randomised controlled trial. Lancet. 2009 Oct 17;374(9698):1351-63. doi: 10.1016/S0140-6736(09)61069-2. Epub 2009 Sep 15. PMID 19762075
- [Background] Ko M, dos Santos PR, Machuca TN, Marseu K, Waddell TK, Keshavjee S, Cypel M. Use of single-cannula venous-venous extracorporeal life support in the management of life-threatening airway obstruction. Ann Thorac Surg. 2015 Mar;99(3):e63-5. doi: 10.1016/j.athoracsur.2014.12.033. PMID 25742860
- [Background] Yusuff HO, Zochios V, Vuylsteke A. Extracorporeal membrane oxygenation in acute massive pulmonary embolism: a systematic review. Perfusion. 2015 Nov;30(8):611-6. doi: 10.1177/0267659115583377. Epub 2015 Apr 24. PMID 25910837
- [Background] Lamhaut L, Jouffroy R, Soldan M, Phillipe P, Deluze T, Jaffry M, Dagron C, Vivien B, Spaulding C, An K, Carli P. Safety and feasibility of prehospital extra corporeal life support implementation by non-surgeons for out-of-hospital refractory cardiac arrest. Resuscitation. 2013 Nov;84(11):1525-9. doi: 10.1016/j.resuscitation.2013.06.003. Epub 2013 Jul 1. PMID 23827888
- [Background] Schmidt M, Hodgson C, Combes A. Extracorporeal gas exchange for acute respiratory failure in adult patients: a systematic review. Crit Care. 2015 Mar 16;19(1):99. doi: 10.1186/s13054-015-0806-z. PMID 25887146
- [Background] Gross-Hardt S, Hesselmann F, Arens J, Steinseifer U, Vercaemst L, Windisch W, Brodie D, Karagiannidis C. Low-flow assessment of current ECMO/ECCO2R rotary blood pumps and the potential effect on hemocompatibility. Crit Care. 2019 Nov 6;23(1):348. doi: 10.1186/s13054-019-2622-3. PMID 31694688
- [Background] Meyer AD, Rishmawi AR, Kamucheka R, Lafleur C, Batchinsky AI, Mackman N, Cap AP. Effect of blood flow on platelets, leukocytes, and extracellular vesicles in thrombosis of simulated neonatal extracorporeal circulation. J Thromb Haemost. 2020 Feb;18(2):399-410. doi: 10.1111/jth.14661. Epub 2019 Nov 14. PMID 31628728
- [Background] Ki KK, Passmore MR, Chan CHH, Malfertheiner MV, Fanning JP, Bouquet M, Millar JE, Fraser JF, Suen JY. Low flow rate alters haemostatic parameters in an ex-vivo extracorporeal membrane oxygenation circuit. Intensive Care Med Exp. 2019 Aug 20;7(1):51. doi: 10.1186/s40635-019-0264-z. PMID 31432279